CLINICAL TRIAL: NCT03815786
Title: XUANRO4 - NATURE 3.1 - Nuovo Approccio Per la Riduzione Delle Tossine Uremiche Renali, REGIONE PUGLIA FSC 2007-2013 Ricerca. Intervento Cluster Tecnologici Regionali
Brief Title: NATURE 3.1_New Approach for the Reduction of REnal Uremic Toxins
Acronym: NATURE31
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XUANRO4-NATURE 3.1
Record Dates: First submitted 2018-11-23; First posted 2019-01-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2018-11

CONDITIONS: Chronic Kidney Diseases; Healthy
Keywords: gut microbiota dysbiosis; uremic toxins; symbiotic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD patients (Experimental): CKD patients stage 3b-4 will follow a 2-months supplementation of either symbiotic or placebo
  Interventions: Dietary Supplement: Symbiotic; Dietary Supplement: Placebo
- Controls (Other): Healthy volunteers will follow a 2-months supplementation of either symbiotic or placebo
  Interventions: Dietary Supplement: Symbiotic; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Symbiotic — 2-months oral administration of the symbiotic supplement (2 bags/day) + 1 month washout
Dietary Supplement: Placebo — 2-months oral administration of the placebo (2 bags/day) + 1 month washout

SUMMARY:
The objective of the pilot study is to validate the clinical use of an innovative symbiotic in patients with chronic kidney disease (CKD) stage 3b-4 and in healthy subjects.

The study aims at evaluating the effects of a symbiotic, consisting of a mixture of probiotics (Lactobacilli and Bifidobacteria), prebiotics (fructooligosaccharides and inulin) and natural antioxidants (a mix of quercetin, resveratrol and proanthocyanidins), by achieving two objectives:

1. Reduction of the serum levels of microbiota-derived uremic toxins, involved in a variety of cardiovascular complications in CKD
2. Reduction of intestinal permeability, inflammatory markers and oxidative stress

ELIGIBILITY:
CKD patients

Inclusion Criteria:

* CKD patients stage 3b-4 not on dialysis
* Aged between 30 to 65
* BMI between 18.5 and 29.9
* Controlled diet
* Informed consent signed

Exclusion Criteria:

* Type 2 diabetes mellitus
* Use of antibiotics or probiotics up to 30 days prior to recruitment
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion or clinical diagnosis of malignancy
* Chronic liver disease
* Treatment with corticosteroids or immunosuppressive drugs
* Previous acute cardiovascular diseases (myocardial infarction, stroke)
* Psychiatric conditions reducing the compliance to treatment protocols

Healthy volunteers

Inclusion Criteria:

* Healthy subjects
* Aged between 35 to 60
* BMI between 18.5 and 29.9
* Medium score of adherence to Mediterranean Diet (PREDIMED score between 6 and 9)
* Informed consent signed

Exclusion Criteria:

* Type 2 diabetes mellitus
* Use of antibiotics or probiotics up to 30 days prior to recruitment
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion or clinical diagnosis of malignancy
* Chronic liver disease
* Treatment with corticosteroids or immunosuppressive drugs
* Previous acute cardiovascular diseases (myocardial infarction, stroke)
* Psychiatric conditions reducing the compliance to treatment protocols

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Change of serum concentration of pCS | 3 months
  Change of p-cresyl sulfate (pCS) serum concentrations assessed by liquid chromatography/mass spectrometry

SECONDARY OUTCOMES:
Change of serum concentration of IS | 3 months
  Change of indoxyl sulfate (IS) serum concentrations assessed by liquid chromatography/mass spectrometry
Change of serum concentration of D-lactate | 3 months
  Change of D-lactate serum concentration (uM)
Change of serum concentration of LPS | 3 months
  Change of lipopolysaccharide (LPS) serum concentration (EU/ml)
Change of percentage of sugar urinary recovery | 3 months
  Change of percentage (%) of urinary recovery of 4 sugars (lactulose, mannitol, sucrose and sucralose)
Change of serum concentration of inflammatory markers | 3 months
  Change of interleukin (IL)6, IL10, IL17, pentraxin3 (PTX3) serum concentrations (pg/ml) evaluated by ELISA
Change of serum concentration of NO | 3 months
  Change of nitric oxide (NO) serum concentration (uM) evaluated by spectrometry

OTHER OUTCOMES:
Gut microbiota | 3 months
  Change of the relative abundance (%) of Operational Taxonomic Units (OTUs) of Firmicutes, Bacteroidetes, Proteobacteria, Verrucomicrobia, Actinobacteria, Synergistetes, Cyanobacteria, Euryarchaeota, Chloroflexi, Nitrospirae, Tenericutes, Fusobacteria, Thermotogae, Acidobacteria evaluated by fecal bacterial DNA genome sequencing.
Change of GI symptoms | 3 months
  Change of gastrointestinal symptoms evaluated by Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire (15 items scored 0-3 each, 0 representing the best and 3 the worse outcome for each item)
Change of stool type | 3 months
  Change of stool type evaluated by BRISTOL Stool Scale (range 1-7, lower and higher values representing worse outcome, middle values representing better outcome)
Change of serum concentration of TMAO | 3 months
  Change of trimethylamine-N-oxide (TMAO) serum concentrations assessed by liquid chromatography/mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari
Locations (1):
- AUO Policlinico Consorziale, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vacca M, Celano G, Calabrese FM, Rocchetti MT, Iacobellis I, Serale N, Calasso M, Gesualdo L, De Angelis M. In vivo evaluation of an innovative synbiotics on stage IIIb-IV chronic kidney disease patients. Front Nutr. 2023 Jun 15;10:1215836. doi: 10.3389/fnut.2023.1215836. eCollection 2023. PMID 37396126